CLINICAL TRIAL: NCT06404060
Title: RECOVER-ENERGIZE: A Platform Protocol for Evaluation of Interventions for Exercise Intolerance in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-ENERGIZE Platform Protocol_Appendix A (Exercise Intolerance)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00112409_A; OT2HL156812 (NIH); NHLBI Grant to RTI (Other Grant/Funding Number: RTI subcontracting with DCRI)
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Long COVID; Long Covid19; Long Covid-19
Keywords: PASC; Exercise; PEM (post exertional malaise)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This platform protocol is designed to allocate participants into an appropriate intervention appendix based on their symptoms of exercise intolerance. Once assigned to an appendix, eligible participants are randomized in a 1:1 ratio to either the study intervention group or a control group.
Who Masked: Outcomes Assessor
Masking Description: The assessor of the primary outcome, Endurance Shuttle Walk Test (ESWT), is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiopulmonary Rehabilitation (Exercise Intolerance) (Experimental): Participants assigned to Cardiopulmonary Rehabilitation will undergo a 12-week personalized cardiopulmonary rehabilitation intervention with a follow-up period of 3 months (total study duration of 6 months).
  Interventions: Behavioral: Personalized Cardiopulmonary Rehabilitation
- Education (Active Comparator): Participants in this group will receive two general education sessions at the start of the intervention with weekly phone/virtual follow-ups from site study staff.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Personalized Cardiopulmonary Rehabilitation — Participants in this group will complete 2-3 cardiopulmonary rehabilitation sessions per week, for 12 weeks, as tolerated. Rehabilitation sessions are provided by respiratory therapists, exercise physiologists, physical therapists, nurses, or others who have experience and training in either pulmonary or cardiac rehabilitation.
  Rehabilitation sessions (adjusted based on the participant's baseline assessment, symptoms, and progress) last about 1 hour and include education, aerobic exercise, strength, and flexibility training.
  Arms: Cardiopulmonary Rehabilitation (Exercise Intolerance)
Other: Education — Participants in this group will receive two general education sessions at the start of the intervention with weekly phone/virtual follow-ups from site study staff.
  Arms: Education

SUMMARY:
This is a platform protocol designed to be flexible so that it is suitable for a range of interventions and settings within diverse health care systems and community settings with incorporation into clinical COVID-19 management programs and treatment plans if results achieve key study outcomes.

This protocol is a prospective, multi-center, multi-arm, randomized, controlled platform trial evaluating interventions to address and improve exercise intolerance and post-exertional malaise (PEM) as manifestations of Post-Acute Sequelae of SARS-CoV-2 Infection (PASC).

The focus of this protocol is to assess interventions that can improve exercise capacity, daily activities tolerance, and quality of life in patients with PASC.

DETAILED DESCRIPTION:
Study interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix. Study intervention appendices may be added or removed according to adaptive design and/or emerging evidence.

The platform protocol enrolls participants who meet study eligibility criteria. After completing initial screening assessments, eligible participants are assigned to one of the study intervention appendices that are actively enrolling. Participants must meet certain criteria within a specific appendix in order to be included in that appendix. Once assigned to an appendix, eligible participants are randomized to either the study intervention group or a control group.

ELIGIBILITY:
Inclusion Criteria:

• See NCT06404047 for RECOVER-ENERGIZE: Platform Protocol level inclusion and exclusion criteria which applies to this appendix

Additional Appendix A (Cardiopulmonary Rehabilitation (Exercise Intolerance)) Level Exclusion Criteria:

1. Known pre-existing postural orthostatic tachycardia syndrome, not related to SARS-CoV-2 infection
2. Known uncontrolled hypertension (blood pressure [BP] ≥ 160/100 mmHg at rest)
3. Any of the following within 4 weeks of enrollment - acute myocardial infarction, unstable angina, uncontrolled arrhythmias causing symptoms or hemodynamic compromise, acute myocarditis or pericarditis, uncontrolled acutely decompensated heart failure (acute pulmonary edema), acute pulmonary embolism, suspected dissecting aneurysm, severe hypoxemia at rest, thromboembolic event(s), any acute or chronic disorder that may affect exercise capacity or be aggravated by exercise (e.g., infection, exercise induced syncope, thyrotoxicosis, unable to cooperate)
4. Score of 2 or greater for both frequency and severity for any of the first 5 questions on the Screening mDSQ-PEM AND answer of 'YES' to either item 7 or 8 on the Screening mDSQ-PEM, and response of > 14 hours in item 9 OR Score of 3 or greater on any severity question (regardless of frequency) AND answer of 'YES' to either item 7 or 8 on the Screening mDSQ-PEM, and response of > 14 hours in item 9 OR Any score of 3 or greater on any of the severity questions on the mDSQ-PEM 48-72 hours following the Screening ISWT test
5. A selection of ≥ 8 on question 1 or ≥ 9 on question 3 of the OH Activity Scale from the mOHQ
6. Engaged in purposeful moderate or greater intensity exercise with the intent to improve one's health 2 or more times per week over the 30 days prior to informed consent
7. Inability to walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Endurance Shuttle Walk Test (ESWT) | Baseline, week 12 (End of Intervention (EOI))
  The ESWT consists of timed walking on a 10m course. The result is expressed as total walking time after an initial 2-minute warm-up. The ESWT is an outcome measure of exercise capacity.
Percentage of participants meeting pre-specified change (minimal important difference) from baseline to End of Intervention on the ESWT | Week 12 (EOI)
  The ESWT consists of timed walking on a 10m course. The result is expressed as total walking time after an initial 2-minute warm-up. The ESWT is an outcome measure of exercise capacity.

SECONDARY OUTCOMES:
Change in physical function, as measured by the PROMIS SF-Physical Function (PROMIS-PF) | Baseline, week 6 (middle of intervention), week 12 (EOI) and week 24 End of Study (EOS)
  The PROMIS Short Form v2.0 - Physical Function 8b (PROMIS-PF) consists of 8 items. The PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities.
Change in physical function, as measured by actigraphy | Baseline, week 6 (middle of intervention), week 12 (EOI) and week 24 End of Study (EOS)
Change in symptom frequency, as measured by the Modified DePaul Symptom Questionnaire - Post-Exertional Malaise (mDSQ-PEM) | Baseline, week 6 (middle of intervention), week 12 (EOI) and week 24 End of Study (EOS)
  Symptom frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time.
Change in symptom severity, as measured by the Modified DePaul Symptom Questionnaire - Post-Exertional Malaise (mDSQ-PEM) | Baseline, week 6 (middle of intervention), week 12 (EOI) and week 24 End of Study (EOS)
  Symptom severity is rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
Change in symptom duration, as measured by the Modified DePaul Symptom Questionnaire - Post-Exertional Malaise (mDSQ-PEM) | Baseline, week 6 (middle of intervention), week 12 (EOI) and week 24 End of Study (EOS)

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Felker, MD, Study Chair — Duke Clinical Research Institute; Barry Make, MD, Study Chair — National Jewish Health; Lucinda Bateman, MD, Study Chair — Bateman Horne Center; Janna Friedly, MD, MPH, Study Chair — University of Washington
Locations (1):
- All sites listed under NCT06404047, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The summary of the results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT06404060/ICF_000.pdf